CLINICAL TRIAL: NCT02869464
Title: The University of Virginia Brain and Aortic Aneurysm Study
Brief Title: UVA Brain and Aortic Aneurysm Study
Acronym: BAAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bradford Worrall, MD, Bradford B. Worrall, M.D., University of Virginia
Other Study IDs: 17341
Record Dates: First submitted 2014-12-01; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Intracranial Aneurysm; Abdominal Aortic Aneurysm
Keywords: Aneurysm; Intracranial Aneurysm; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aortic Aneurysm, Abdominal; Aneurysm | interventions — High-Energy Shock Waves; DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Approximately 3 mL of blood are obtained via venipuncture at the time of subject consent for banking and future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients presenting with IA: These patients will undergo an abdominal ultrasound (Imaging - Ultrasound) to test for abdominal aortic aneurysm(s). RNA, DNA testing will be planned on banked samples
  Interventions: Other: Imaging-Ultrasound; Genetic: DNA, RNA testing
- Patients presenting with AAA: These patients will undergo a non-contrast enhanced magnetic resonance angiogram (MRA) (Imaging - MRA) to test for intracranial aneurysm(s). RNA, DNA testing will be planned on banked samples
  Interventions: Other: Imaging-MRA; Genetic: DNA, RNA testing

INTERVENTIONS:
Other: Imaging-Ultrasound — Abdominal Ultrasound
  Groups: Patients presenting with IA
Other: Imaging-MRA — Non-contrast Enhanced Magnetic Resonance Angiogram
  Groups: Patients presenting with AAA
Genetic: DNA, RNA testing — To test for the co-prevalence of shared genetic markers in afflicted populations.

SUMMARY:
The purpose of this study is to examine the percentage of patients who present with abdominal aortic aneurysms (AAA) will also have intracranial aneurysms (IA) and conversely; to examine the percentage of patients who present with intracranial aneurysms will also have abdominal aortic aneurysms.

DETAILED DESCRIPTION:
The investigators have previously generated estimates for cost effectiveness of each arm of this reciprocal screening protocol based on literature dervied estimates of coprevalence and other key factors in a decision tree model to compare costs and outcomes. They measured expected outcomes using quality-adjusted life years (QALY) and the incremental cost-effectiveness ratios (ICER). The current study will involve establishment of the true co-prevalence and recalculation of the ICERs and QALYs. Based on their literature derived models we previously found an ICER of $34.01/QALY for AAA screening in IA patients and an ICER of $6,401.91/QALY for IA screening in AAA patients. Both of these are well below the societal accepted threshold of $60,000/QALY. However, both models were sensitive to co-prevalence. In the current study the investigators will therefore determine the actual cost-effectiveness of performing additional radiographic procedures and genetic counseling. The investigators will also bank DNA and RNA for future research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical and radiographic diagnosis of either abdominal aortic aneurysm (AAA) or intracranial cerebral aneurysm (IA). Aneurysm may be symptomatic (s/p rupture or mass effect) or asymptomatic (detected as part of screening or incidentally discovered. Aneurysms int he brain may be multiple. AAA will be defined as >= 3 cm by any imaging modality. IA will be defined as >= 3 mm on any imaging modality.
* Able to provide a valid informed consent (self or legally authorized representative)

Exclusion Criteria:

* Contra-indication for MRI/A (embedded metal, intractable claustrophobia, pacemaker, etc.)
* Intracranial aneurysm associated with arteriovenous malformation
* Clinical or radiographic diagnosis of mycotic aneurysm
* Substantial pre-existing neurological or psychiatric illness that would confound neurological assessment or other outcome assessment.
* Other serious conditions that make the patient unlikely to survive long enough to benefit from the screening program.
* Inability to follow the protocol or return for screening test or genetic counseling.
* Unwilling to have reports from imaging and genetic counselor sent to a clinician (PCP, testing surgeon, etc)

Note: Pregnancy is not a reason to exclude, but imaging done for the study will be postponed until after the subject has given birth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with either a IA or AAA.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Revised cost-effective analysis measured in dollars/quality adjusted life years (QALY) | 2 years
  Revision of cost effective analysis for screening for AAA in those presenting with IA and for screening for IA in those with AAA.

SECONDARY OUTCOMES:
Analysis of Covariates for co-prevalence of aneurysms measured as present or absent | Year 2
  Analysis of covariates associated with co-prevalence of aneurysms in both territories.
Biorepository (samples stored in freezer) | Year 2
  Develop a biorepository of DNA and RNA for individuals presenting with either IA or AAA, allowing specific future testing of shared genetic risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Bradford B Worrall, MD, MSc, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Summary data will be shared and published.